CLINICAL TRIAL: NCT03134885
Title: Evaluation of a Regional Post-discharge Monitoring System for Suicide Attempters in the North-Pas de Calais Region of France
Brief Title: Evaluation of a Regional Post-discharge Monitoring System for Suicide Attempters
Acronym: EVAL-VIGILANS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Regional Agency of Sante Nord Pas-de-Calais (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_52; 2015-A01984-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-04-13; First posted 2017-05-01 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2021-04

CONDITIONS: Suicide, Attempted
Keywords: suicide; suicidal conducts; post discharge monitoring system
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VigilanS Nord-Pas de Calais cohort: All patients leaving in the Nord-Pas de Calais region and entering in the VigilanS program after a suicide attempt

SUMMARY:
VigilanS is an innovative healthcare program. Participants of this program are all patients leaving in the Nord-Pas de Calais region who survived a suicide attempt.

General goals of the post hospitalization monitoring system for suicidal attempters are:

* Standardize general healthcare's practices by offering alert networks and innovative response procedures in case of suicidal crisis.
* Coordinate the various health partners' actions around the patient (GP, psychiatrist, psychologist).
* Contribute to reducing mortality and morbidity by suicide (subsequent suicide) in determined territories.

The evaluation of VigilanS will be quantitative and qualitative.

DETAILED DESCRIPTION:
Every patient who is discharged after a suicidal gesture will be proposed to enter the program. He will be handed a "green card" with a toll-free and unique phone number and an information letter which explains the program and his rights as a patient.

Phone calls Calling team is composed of 4 psychologists and 3 psychiatric nurses especially trained to detect and manage suicidal crises. Monday to Friday, from 9 AM until 6 PM, there is two callers located in the emergencies' calling center. They will give calls to patients after their entry in the program and they will also receive incoming calls at the number available on "green cards" handed to patients.

Calls 10 days after discharge

Subjects who did at least two suicidal attempts before entering the VigilanS program will be call 10 to 20 days after their discharge from the hospital.

After every call, a short report is sent to the patient psychiatrist or his GP. 6 months calls

For every suicide attempters included in the program, a call is planned at the end of the sixth month after discharge from the hospital. This call aims to make a clinical review of patient and propose the end of the monitoring. If needed, the monitoring program can be reset for a 6 months period. In order to structure the call and gather data on the program evaluation, the six months call includes a psychological assessment by Mini International Neuropsychiatric Interview / MINI DSM V (Sheehan et al. 1998) and by the Columbia Suicide Severity rating Scale C-SSRS (Posner et al. 2011) as well as a global satisfactory survey on the program. If a contacted subject represents a high suicide risk, callers can trigger various actions like in a 10 days call.

If patient is unreachable a unique postcard will be sent to remind him of VigilanS coordinates. After every call, a short report is sent to the patient psychiatrist or his GP.

Postcards After every contact, but mostly after a 10 days call, the caller can decide to send 4 personalized post cards to a patient. One postcard is sent by month on a period of four months. Cards are embodied by patient name, logo of the structure which included him and coordinates of including department.

Quantitative evaluation will assess:

* Profiles of patients with good respond to the program or not (who had or not attempted suicide within 6 months)
* Development of partnership within the program (number of facilities sharing the system, number of patients in the program compared to overall number of suicide attempters addressed to one centre…).
* Program efficiency "in real life" on reduction of suicidal conducts. Using four comparator tools :

  * Evolution of suicidal conducts since the implementation of VigilanS in a specific center (comparison "before / after").
  * Evolution of suicidal conducts between a region implementing VigilanS and a region which doesn't, upon the same period of time (comparison "here/there").
  * Comparison of subsequent suicide attempts rate between patients in VigilanS and patients benefiting of "treatment as usual", within a year.
  * Comparison of mortality by suicide rate.
* The impact of VigilanS on a patient's care pathway based on data from CNAMTS' database (National health insurance system).

Qualitative evaluation will assess the system acceptability by patients and professionals and also the variation of representations of suicide by different professionals which are in contact with suicidal patients.

ELIGIBILITY:
Inclusion Criteria:

* leaving in the Nord-Pas de Calais region
* entering in the VigilanS program after a suicide attempt

Exclusion Criteria:

* refusal to enter in the program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients leaving in the Nord-Pas de Calais region who survived a suicide attempt and entering in the VigilanS program when they discharge from the hospital
Sampling Method: Non-Probability Sample
Enrollment: 12989 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
If patients had or not attempted suicide | 6 months
  Yes or no
Sex | 6 months
Age | inclusion
Marital status | inclusion
Means of suicide attempts | 6 months
Reason of suicide attempts | 6 months
Length of the hospital stay at inclusion | inclusion
Presence of accompanying people | inclusion
MINI (Mini International Neuropsychiatric Interview) lifetime 5.5.0 | 6 months
  psychopathological evaluation
Columbia Suicide Severity Rating Scale C-SSRS | 6 months
  review of suicidal behaviours and thoughts
Number of emergency calls | 6 months
Number of subsequent suicide attempts | 6 months
Number of hospitalization after a suicide attempt | 6 months

SECONDARY OUTCOMES:
Number of suicidal attempts in Nord-Pas de Calais region | each year during 3 years
Local mortality by suicide | each year during 3 years
Number of suicidal conducts in Picardie region | 1 year
Number of hospital stays after a suicide attempt | each year during 3 years
  Obtained from PMSI's data (French register of hospitals economics management)
Care pathway | 1 year
  GP or psychiatrist appointments, medical treatment, and hospitalization in psychiatric facility : with CNAM (National health insurance system) data
Number of "green cards" distributed | each year during 3 years
Number of incoming and outgoing calls | each year during 3 years
Number of phone intervention and of calls leading to triggering of emergency department | each year during 3 years
Number of postcards sent | each year during 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Vaiva, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (28):
- France (28):
  - General Hospital, Armentieres, Armentières
  - General Hospital, Arras, Arras
  - General Hospital, Bethune, Béthune
  - General Hospital, Boulogne sur Mer, Boulogne-sur-Mer
  - General Hospital, Calais, Calais
  - General Hospital, Cambrai, Cambrai
  - General Hospital, Denain, Denain
  - General Hospital, Douai, Douai
  - General Hospital, Dunkerque, Dunkirk
  - General Hospital, Fourmies, Fourmies
  - General Hospital, Hazebrouck, Hazebrouck
  - Clinic Fleury, Hénin Beaumont, Hénin-Beaumont
  - Polyclinic, Henin-Beaumont, Hénin-Beaumont
  - General Hospital, Lens, Lens
  - Riaumont's Polyclinic, Liévin, Liévin
  - St Vincent's Hospital, Lille, Lille
  - University Hospital, Lille, Lille
  - St Philibert's Hospital, Lomme, Lomme
  - Genral Hospital, Maubeuge, Maubeuge
  - General Hospital, Montreuil sur Mer, Montreuil-sur-Mer
  - General Hospital, Roubaix, Roubaix
  - Lucien Bonnafé Hospital, Roubaix, Roubaix
  - General Hospital, St Omer, Saint-Omer
  - EPSM, St Venant, Saint-Venant
  - General Hospital, Seclin, Seclin
  - EPSM, Tourcoing, Tourcoing
  - General Hospital, Tourcoing, Tourcoing
  - General Hospital, Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demesmaeker A, Creupelandt C, Leroy A, Vaiva G, D'Hondt F. Impact of posttraumatic stress disorder and comorbid psychiatric conditions on suicide reattempts. Eur J Psychotraumatol. 2025 Dec;16(1):2461435. doi: 10.1080/20008066.2025.2461435. Epub 2025 Feb 12. PMID 39936356
- [Derived] Demesmaeker A, Amad A, Chazard E, Demarty AL, Schlienger H, Lehmann E, Debien C, Jardon V, Bounebache K, Rey G, Vaiva G. Suicide and All-Cause Mortality Within 1 Year After a Suicide Attempt in the VigilanS Cohort. J Clin Psychiatry. 2023 Sep 11;84(6):22m14520. doi: 10.4088/JCP.22m14520. PMID 37707316
- [Derived] Fossi LD, Debien C, Demarty AL, Vaiva G, Messiah A. Suicide reattempt in a population-wide brief contact intervention to prevent suicide attempts: The VigilanS program, France. Eur Psychiatry. 2021 Jul 16;64(1):e57. doi: 10.1192/j.eurpsy.2021.2221. PMID 34266505
- [Derived] Duhem S, Berrouiguet S, Debien C, Ducrocq F, Demarty AL, Messiah A, Courtet P, Jehel L, Thomas P, Deplanque D, Danel T, Walter M, Notredame CE, Vaiva G. Combining brief contact interventions (BCI) into a decision-making algorithm to reduce suicide reattempt: the VigilanS study protocol. BMJ Open. 2018 Oct 23;8(10):e022762. doi: 10.1136/bmjopen-2018-022762. PMID 30355792